CLINICAL TRIAL: NCT03388047
Title: Prospective Pilot Cohort Study to Assess Feasibility of Multi-Spectral Endoscopic Imaging for Detection of Early Neoplasia in Barrett's Oesophagus
Brief Title: Feasibility of Multi-Spectral Endoscopic Imaging for Detection of Early Neoplasia in Barrett's Oesophagus
Acronym: MuSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Principal Investigator, Honorary Gastroenterology Consultant, University of Cambridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MuSE version 1
Record Dates: First submitted 2017-11-23; First posted 2018-01-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Barrett Esophagus; Esophageal Neoplasms; Reflux Esophagitis
Keywords: Barrett Esophagus; Endoscopy; Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Esophagitis, Peptic; Adenocarcinoma | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Barrett's Esophagus patients (Experimental): Multi-Spectral Endoscopic Imaging
  Interventions: Device: Endoscopy with Polyscope (Polydiagnost TM) coupled with Multi-Spectral Imaging light-source

INTERVENTIONS:
Device: Endoscopy with Polyscope (Polydiagnost TM) coupled with Multi-Spectral Imaging light-source — During surveillance endoscopy procedure, the endoscopist will insert the multispectral endoscopy probe through the working channel and use this to inspect the Barrett's oesophagus segment and any visible lesions

SUMMARY:
Multispectral imaging represents an exciting new field of investigation in endoscopic research. Multispectral imaging uses a specialised camera to detect multiple colours, allowing us to build a rough spectrum from each point in our image. It is widely reported that these spectra are different for different tissue types, but this is difficult to study ex vivo since de-oxygenation of the blood and decay of the tissue change these spectra considerably.

The investigators have therefore designed this study to asses the different multispectral imaging spectra of Barrett's Oesophagus, which we believe might be utilised as a method to detect dysplasia in the future.

DETAILED DESCRIPTION:
The investigators have developed a custom multispectral endoscopes based around a CE marked device, the PolyScope disposable endoscope (PolyDiagnost). This is a combined sterile catheter and fibre optic device designed to optimize light delivery to the anatomy and to acquire and transmit endoscopic images back to a camera. This CE marked system can be used to endoscope luminal organs such as the oesophagus, but also biliary tract, the bladder and the oro-pharynx.

The PolyScope can be inserted thought the accessory channel of commercial endoscopes. The design of the fibre optic device is durable and re-useable; it is inserted within the disposable sterile catheter channel, which is able to flex and bend to orient the device to the region of interest for imaging. The fibre optic device never comes into contact with the patient. The sterile catheter, which shields the fibre optic device, is disposed following a procedure.

The use of the PolyScope provides the advantage of building on a known system. The commercial PolyScope probe is coupled outside of the patient to a custom multispectral detection and illumination system. No modified part of the device comes into contact with the patient.

The patients recruited to this study will have a clinical indication to an endoscopic examination for Barrett's oesophagus or early oesophageal adenocarcinoma. There will not be extra procedures involved. The experimental part of the procedure, using Polyscope multispectral endoscope will prolong the procedure in most cases by approximately 5-10 minutes

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over 18 years
* Previous diagnosis of Barrett's oesophagus, with an endoscopic length of at least 2 cm
* Previous diagnosis of oesophageal glandular dysplasia or early oesophageal adenocarcinoma for consideration of endoscopic therapy

Exclusion Criteria:

* History of oesophageal stricture precluding passage of the endoscope,
* Pregnancy, or planned pregnancy during the course of the study,
* Currently breastfeeding
* Any history of esophageal varices, liver impairment of moderate or worse severity (Child's- Pugh class B & C) or evidence of varices on initial treatment endoscopy,
* Any history of oesophageal surgery, except for uncomplicated fundoplication, and,
* History of coagulopathy, with INR>1.3 and/or platelet count of <75,000.
* On clopidogrel, and/or warfarin for high risk condition and unable to withhold temporarily the medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Level of confidence in delineating the area of interest by multispectral imaging | 1 year
  Level of confidence in delineating the area of interest by the multispectral endoscope in terms of image quality and visibility of area of interest assessed by endoscopist using a 1 to 10 Visual Analogue Score (VAS). We will consider the following ranges 0-3 poor; 4-5 fair; 6-8 good, 9-10 excellent

SECONDARY OUTCOMES:
Imaging spectra by multispectral endoscopy in neoplastic vs. non-neoplastic Barrett's | 1 year
  Number and type of image spectra corresponding to neoplastic and non-neoplastic area of Barrett's Oesophagus
Patient comfort | 1 year
  Patient comfort score measured by assisting nurse according to standard scoring scale (1 to 5)
Time | 1 year
  Time to perform multispectral imaging in minutes
Correlation with molecular biomarkers | 1 year
  Comparison of the biomarker features of biopsies directed by multispectral imaging (both neoplastic and non-neoplastic) using a molecular panel assessing aneuploidy, p53 and cyclin A.

CONTACTS AND LOCATIONS:
Locations (1):
- MRC Cancer Unit, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waterhouse DJ, Bano S, Januszewicz W, Stoyanov D, Fitzgerald RC, di Pietro M, Bohndiek SE. First-in-human pilot study of snapshot multispectral endoscopy for early detection of Barrett's-related neoplasia. J Biomed Opt. 2021 Oct;26(10):106002. doi: 10.1117/1.JBO.26.10.106002. PMID 34628734